CLINICAL TRIAL: NCT07106736
Title: A Prospective, Open-Label, Single-Center Clinical Study of a Fully Immunotherapy-Based Strategy Driven by MRD-Guided Dynamic Risk Stratification in Transplant-Ineligible Newly Diagnosed Multiple Myeloma
Brief Title: MRD-Adaptive Guided Immunotherapy With CAR-T for Transplant-Ineligible Patients With Multiple Myeloma
Acronym: MAGIC-TIEMM
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IIT2025064
Record Dates: First submitted 2025-07-30; First posted 2025-08-06 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-07

CONDITIONS: Multiple Myeloma, Newly Diagnosed
Keywords: Multiple myeloma; MRD; CAR-T; BiTEs
MeSH Terms: conditions — Multiple Myeloma; Bites and Stings

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard-risk (Experimental): Enrolled patients will be stratified into standard-risk group based on the absence of ultra-high-risk features, defined as: (1) double-hit cytogenetics, (2) presence of extramedullary disease, or (3) circulating tumor cells (CTCs) ≥2%. Patients in the standard-risk group will receive BCMA CAR-T therapy after standard induction, followed by standard consolidation and maintenance. Patients achieving sustained MRD negativity and stringent complete response (sCR) on two consecutive assessments may enter a treatment-free observation phase. Patients who experience MRD resurgence or loss of response will resume maintenance therapy.
  Interventions: Biological: BCMA CAR-T
- Ultra high risk (Experimental): Enrolled patients will be stratified into an ultra-high-risk group based on the presence of ultra-high-risk features, defined as: (1) double-hit cytogenetics, (2) presence of extramedullary disease, or (3) circulating tumor cells (CTCs) ≥2%. Patients in the ultra-high-risk group will also receive BCMA CAR-T therapy after induction, followed by GPRC5D/CD3 bispecific antibody consolidation and maintenance. Patients achieving sCR and sustained MRD negativity (≥12 months) may enter treatment-free observation, while those with MRD resurgence or loss of response will resume maintenance therapy.
  Interventions: Biological: BCMA CAR-T; Drug: GPRC5D/CD3 BiTEs

INTERVENTIONS:
Biological: BCMA CAR-T — Patients will receive single-dose infusion of autologous BCMA-directed CAR-T cellsBCMA CAR-T single dose (3.0 x 10^6 cells /kg).
Drug: GPRC5D/CD3 BiTEs — Patients will receive GPRC5D/CD3 BiTEs maintenance therapy at a dose of 54 μg/kg every 4 weeks, starting 3 months after BCMA CAR-T infusion.
  Arms: Ultra high risk

SUMMARY:
This is a prospective, single-center, clinical study to evaluate the efficacy and safety of a fully immunotherapy-based strategy guided by MRD-driven dynamic risk stratification in transplant-ineligible patients with newly diagnosed multiple myeloma.

DETAILED DESCRIPTION:
All subjects will receive standard induction therapy for up to four cycles prior to screening. Following response evaluation, those who meet the inclusion criteria will be enrolled and subsequently stratified into standard-risk and ultra-high-risk groups based on predefined clinical and molecular features.

Patients in the standard-risk group will receive BCMA CAR-T therapy, followed by standard consolidation and maintenance. Patients achieving sustained MRD negativity and stringent complete response (sCR) on two consecutive assessments may enter a treatment-free observation phase. Patients in the ultra-high-risk group will also receive BCMA CAR-T therapy, followed by GPRC5D/CD3 bispecific antibody consolidation and maintenance. Patients achieving sCR and sustained MRD negativity (≥12 months) may enter treatment-free observation. Patients who experience MRD resurgence or loss of response will resume maintenance therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years and ≤ 75 years.
2. Participants with documented newly-diagnosed multiple myeloma according to IMWG diagnostic criteria.
3. Measurable disease at screening, defined as: Serum M-protein level ≥1.0 g/dL or urine M-protein level ≥200 mg/24 hours; or Light chain MM without measurable disease in serum or urine: serum Ig free-light chain (FLC) ≥10 mg/dL and abnormal serum Ig kappa lambda FLC ratio.
4. Patients deemed ineligible for high-dose chemotherapy with ASCT due to any of the following: Age ≥65 years; Investigator assessment of ineligibility; ECOG performance status 3-4; Repeated failure of hematopoietic stem cell mobilization; Patient's decision to defer ASCT.
5. Tumor cells were BCMA and GPRC5D positive.
6. Serum total bilirubin <2 x upper limit of normal (ULN), serum AST and ALT <3 x ULN, creatinine clearance ≥ 30mL/min (Cockroft-Gault formula).
7. Informed Consent/Assent: All subjects have the ability to understand and the willingness to sign a written informed consent.

Exclusion Criteria:

1. Active amyloidosis.
2. Central nervous system involvement.
3. Prior BCMA-targeted therapy or CAR-T therapy.
4. Active hepatitis B or hepatitis C virus infection.
5. Known HIV infection.
6. Life expectancy <6 months.
7. Woman who are pregnant or breastfeeding.
8. Evidence of uncontrolled dysfunction of heart, lung, brain, and other important organs.
9. Any other conditions that are not eligible for the trial in the judgement of the principal investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-08-10 (Estimated); Primary Completion 2027-08-01 (Estimated); Study Completion 2029-08-01 (Estimated)

PRIMARY OUTCOMES:
Sustained MRD-negative rate | Up to 2 year
  Rate of patients achieving sustained MRD negativity for more than 12 months
Progression free survival (PFS) | Up to 3 year
  Progression free survival is defined as the time from the date of diagnosis to the date of first documented PD, as defined in the IMWG criteria, or death due to any cause, whichever occurs first

SECONDARY OUTCOMES:
Complete response rate (CRR) | Up to 2 years
  CR or better is defined as percentage of participants who achieve a CR response or Stringent Complete Response (sCR) response accoording to the IMWG criteria.
MRD negativity rate | Up to 2 years
  Rate of patients achieving MRD negativity
Overall survival (OS) | Up to 5 year
  Overall survival is defined as the time from the date of diagnosis to the date of death due to any cause

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Hematology and Blood Diseases Hospital Chinese Academy of Medical Sciences, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: No